CLINICAL TRIAL: NCT04135833
Title: A Phase I Study to Assess the Effect of Itraconazole and Rifampicin on Pharmacokinetics Profile of BPI-7711 in Chinese Healthy Volunteers
Brief Title: A Phase I Study to Assess the Effect of Itraconazole and Rifampicin on Pharmacokinetics Profile of BPI-7711
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beta Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BPI-7711DDI
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: NSCLC
MeSH Terms: interventions — rezivertinib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole and BPI-7711 (Experimental): BPI-7711 alone followed by BPI-7711 +Itraconazole, followed by Itraconazole alone.
  Interventions: Drug: BPI-7711; Drug: Itraconazole
- Rifampicin and BPI-7711 (Experimental): BPI-7711 alone followed by BPI-7711 +Rifampicin, followed by Rifampicin alone.
  Interventions: Drug: BPI-7711; Drug: Rifampicin

INTERVENTIONS:
Drug: BPI-7711 — BPI-7711 60 mg
  Other Names: BPI-7711 capsule
  Arms: Itraconazole and BPI-7711
Drug: BPI-7711 — BPI-7711 180 mg
  Other Names: BPI-7711 capsule
  Arms: Rifampicin and BPI-7711
Drug: Itraconazole — Itraconazole 200 mg
  Other Names: Itraconazole capsule
  Arms: Itraconazole and BPI-7711
Drug: Rifampicin — Rifampicin 600 mg
  Other Names: Rifampicin capsule
  Arms: Rifampicin and BPI-7711

SUMMARY:
This is a phase I study to assess the effect of itraconazole and rifampicin on the pharmacokinetic parameters of BPI-7711 in Chinese healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged from 18 to 45 years
* BMI from 18.5 to 28.0 kg/m2
* Medical history, vital signs, physical examination and lab tests are normal or abnormal without clinical significance

Exclusion Criteria:

* Subjects with clinical significant diseases
* Subjects with allergic disease history
* Subjects with gastrointestinal disease history that can affect study drug absorption
* Subjects with drug abuse history

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples collected on Day 1 and Day 20 (arm 1)/Day 25 (arm 2) at pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168 and 336 hours post BPI-7711 dose
  Pharmacokinetics of BPI-7711 by assessment of maximum plasma concentration
AUC(0-last) | Blood samples collected on Day 1 and Day 20 (arm 1)/Day 25 (arm 2) at pre-dose, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168 and 336 hours post BPI-7711 dose
  Pharmacokinetics of BPI-7711 by assessment of area under the plasma concentration time curve from zero to last assessed timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No